CLINICAL TRIAL: NCT06749340
Title: Examination of the Effects of Face-to-Face and Home-Based Resistive Exercise Program on Muscle Strength, Muscle Mass and Cognitive Functions in Individuals with Compensated Liver Cirrhosis: Randomized Controlled Single -Blind Study
Brief Title: Examining the Effects of Different Resistive Exercise Programs in Individuals with Compensated Liver Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Mustafa Oğuz Kethudaoglu, Pirincipal Investigator; PT, MSc, PhD (c), Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-6055 / 927
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Coginitive Dysfunction; Compensated Liver Cirrhosis; Physical Dysfunction; Sarcopenia
Keywords: cirrhosis; cognitive dysfunction; sarcopenia; strengthening; telerehabilitation
MeSH Terms: conditions — Sarcopenia; Fibrosis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants with liver cirrhosis will be randomly assigned to 3 groups: face-to-face exercise group, home-based exercise group and control group.
Who Masked: Outcomes Assessor
Masking Description: After the first evaluation, participants will determine their groups by choosing closed and opaque envelopes. One of the researchers will perform all outcome measurements and will not know which group the participant falls into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Face-to-face Exercise Group (Experimental): Participants will undergo exercise sessions 3 days a week for 12 weeks. Sessions will include a warm-up, upper and lower extremity strengthening (1/3 set - 8/12 repetitions) and cool-down program. Theraband will be used in strengthening exercises. Theraband offers different resistance levels with its different colors. In order from lightest to heaviest; skin color, yellow, red, green, blue, black, grey, gold. Exercises (theraband color, intensity, number of sets and repetitions) will be made into a personalized program according to the tolerance level of the participants in the first session. Exercise intensity will be determined using the OMNI - Resistance Exercise Scale (OMNI - RES). The warm-up and cool-down periods in the exercise program will be carried out at levels 9 - 12 according to the Borg Scale.
  Interventions: Other: Assigned Interventions; Other: Face-to-face Exercise
- Home-based Exercise Group (Experimental): Participants will follow the same program as in the face-to-face exercise group. The first meeting with the participants will be held face to face and the details of the study will be explained. Home-based exercises will be carried out with the Fiziu (Fiziu Sağlık Hizmetleri Teknoloji A.Ş., Istanbul, Türkiye) program and the exercise program will be delivered to the participants through this program. Therabands with which the participants will do their exercises will be provided by the researchers. The progression program will be determined in line with the difficulty and effort felt by the participants through weekly meetings.
  Interventions: Other: Assigned Interventions; Other: Home-based Exercise
- Control Group (Other): Participants assigned to the control group will have the same evaluation sessions as participants assigned to the experimental groups. The first evaluation will be made at the beginning of the study, the second evaluation after the 8-week period, the third evaluation after the 12-week period, the fourth evaluation after the 6-month follow-up, and the fifth evaluation after the 12-month follow-up. Participants who will not be included in any study sessions during this process will be included in the study program that appears to be effective as a result of the study. Participants in this group will be offered the program recommended by the US Office of Disease Prevention and Health Promotion and used in individuals who have previously had a liver transplant. This program consists of aerobic exercises (walking, cycling, etc.) starting from 60-65% of the maximum heart rate and progressing to 75-80%.
  Interventions: Other: Assigned Interventions; Other: Control

INTERVENTIONS:
Other: Assigned Interventions — Psychometric Hepatic Encephalopathy Scoring (PHES) Test
  * Digit Symbol Test
  * Number Combination Test-A
  * Number Combination Test-B
  * Serial Punctuation Test
  * Line Drawing Test
    6 Minute Walk Test
    5 Times Sit and Stand Test
  Manual Muscle Test
  Hand Grip Strength Test
  Quadriceps muscle thickness measurement with ultrasonography
  All evaluations will be repeated 5 times.
Other: Face-to-face Exercise — Participants will undergo exercise sessions 3 days a week for 12 weeks. Sessions will include a warm-up, upper and lower extremity strengthening (1/3 set - 8/12 repetitions) and cool-down program. Theraband will be used in strengthening exercises. Theraband offers different resistance levels with its different colors. In order from lightest to heaviest; skin color, yellow, red, green, blue, black, grey, gold. Exercises (theraband color, intensity, number of sets and repetitions) will be made into a personalized program according to the tolerance level of the participants in the first session. Exercise intensity will be determined using the OMNI - Resistance Exercise Scale (OMNI - RES). The warm-up and cool-down periods in the exercise program will be carried out at levels 9 - 12 according to the Borg Scale.
  Arms: Face-to-face Exercise Group
Other: Home-based Exercise — Participants will follow the same program as in the face-to-face exercise group. The first meeting with the participants will be held face to face and the details of the study will be explained. Home-based exercises will be carried out with the Fiziu (Fiziu Sağlık Hizmetleri Teknoloji A.Ş., Istanbul, Türkiye) program and the exercise program will be delivered to the participants through this program. Therabands with which the participants will do their exercises will be provided by the researchers. The progression program will be determined in line with the difficulty and effort felt by the participants through weekly meetings.
  Arms: Home-based Exercise Group
Other: Control — Participants assigned to the control group will have the same evaluation sessions as participants assigned to the experimental groups. The first evaluation will be made at the beginning of the study, the second evaluation after the 8-week period, the third evaluation after the 12-week period, the fourth evaluation after the 6-month follow-up, and the fifth evaluation after the 12-month follow-up. Participants who will not be included in any study sessions during this process will be included in the study program that appears to be effective as a result of the study. Participants in this group will be offered the program recommended by the US Office of Disease Prevention and Health Promotion and used in individuals who have previously had a liver transplant. This program consists of aerobic exercises (walking, cycling, etc.) starting from 60-65% of the maximum heart rate and progressing to 75-80%.
  Arms: Control Group

SUMMARY:
Reasons such as sleep disorders, depression, decreased independence in daily living activities and decreased quality of life, which are seen in the majority of liver cirrhosis patients, can cause cognitive dysfunction, especially attention. It is known that physical dysfunctions are observed in patients with liver cirrhosis along with cognitive dysfunction. Sarcopenia is the most important of these dysfunctions. Sarcopenia is the progressive, widespread loss of muscle mass, function and strength. The aim of this study is to determine the effects of face-to-face and home-based progressive strengthening exercise program performed 3 times a week for 12 weeks on muscle strength, muscle mass, functionality and cognitive functions in individuals with liver cirrhosis. It is also aimed to test the feasibility and effectiveness of the home-based exercise method in individuals with liver cirrhosis. Another aim of our study is to determine the exercise dose required to improve muscle strength, muscle mass, functionality and cognitive functions in individuals with liver cirrhosis and the duration of treatment effectiveness through follow-up.

DETAILED DESCRIPTION:
Reasons such as sleep disorders, depression, decreased independence in daily living activities and decreased quality of life, which are seen in the majority of liver cirrhosis patients, can cause cognitive dysfunction, especially attention. And also, the most typical finding of hepatic encephalopathy is cognitive dysfunction. It is known that hepatic encephalopathy impairs attention, orientation, coordination abilities and slows down information processing processes. It is known that physical dysfunctions are observed in patients with liver cirrhosis along with cognitive dysfunction. Sarcopenia is the most important of these dysfunctions. Sarcopenia is the progressive, widespread loss of muscle mass, function and strength. The European Working Group on Sarcopenia in Older People defined sarcopenia in 2010 as a syndrome characterized by progressive and widespread loss of muscle mass and strength, associated with risks such as physical disability, low quality of life, and death. The rate of sarcopenia development in individuals with liver cirrhosis is around 70%. Sarcopenia has been described primarily in association with old age. Sarcopenia seen in cirrhosis is classified as secondary sarcopenia associated with disease, insufficient physical activity or malnutrition. Exercise may be the most effective intervention for sarcopenic individuals. It is well known that exercise has a positive effect on muscle mass, muscle strength and physical performance. And also, exercise has been proven to be effective in improving cognitive functions, which can improve mental state such as depression and insomnia stress. The aim of this study is to determine the effects of face-to-face and home-based progressive strengthening exercise program performed 3 times a week for 12 weeks on muscle strength, muscle mass, functionality and cognitive functions in individuals with liver cirrhosis. It is also aimed to test the feasibility and effectiveness of the home-based exercise method in individuals with liver cirrhosis. Another aim of our study is to determine the exercise dose required to improve muscle strength, muscle mass, functionality and cognitive functions in individuals with liver cirrhosis and the duration of treatment effectiveness through follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40 and 65;
* Being diagnosed with liver cirrhosis;
* Not having had a liver transplant;
* Being cooperative;
* Volunteering to participate in the study;
* Having a smart device (phone/tablet/computer);
* Having internet access;
* Modified Child-Turcotte-Pugh Score to be A and B.

Exclusion Criteria:

* Having a disease that may affect cognitive functions;
* Having an orthopedic, neurological, psychological, cardiac, renal or pulmonary disease;
* Having a physical or mental disability;
* Having a communication problem;
* Being unable to read or write;
* Modified Child-Turcotte-Pugh Score to be C.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-23 (Estimated); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Cognitive Dysfunction Evaluation - Digit Symbol Test | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  DST is a neurophysiological test that is sensitive to brain damage, dementia and depression. It consists of a table and a list of numbers, with a symbol corresponding to each number. Under each number there is a box where the symbol corresponding to that number will be drawn. The aim is to draw as many symbols correctly as possible in the allotted time. The participant is given the page containing the digit symbol test and the following is said to the participant: "In this test, you will be shown numbers from 1 to 9 and 9 shapes corresponding to each number. We want you to draw the shape under each number in the empty box under the numbers in the table below. First, you will be asked to fill in a line for practice purposes, and then the same process will be done by keeping time. Our goal is to see how many boxes you can fill in 90 seconds." The number of symbols drawn correctly by the participant at the end of the given time is recorded.
Cognitive Dysfunction Evaluation - Number Combination Test-A | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  NCT-A is a test that measures conscious motor ability. NCT-A measures visuospatial orientation and psychomotor speed. The patient is given two pages of NCT-A, first with the practice test and then with the actual test. "In this test, what you are asked to do is to combine the mixed numbers from 1 to 25 by drawing a line with a pencil in numerical order. The point you need to pay attention to while doing this is not to raise your hand and skip the number sequence while drawing." Then the test begins. There is no time keeping in the practice test. Afterwards, it is recorded how long it took to complete the second test.
Cognitive Dysfunction Evaluation - Number Combination Test-B | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  In addition to NCT-A, NCT-B also evaluates the ability to sustain attention. The participant is given the page containing the NCT-B test. "In this test, similar to the NCT-A test, there are numbers from 1 to 13 and letters from A to I. What you are asked to do is to combine the mixed numbers and letters with lines in the form of one number and one letter. The point you need to pay attention to while doing this is not to raise your hand while drawing and not to skip the number-letter sequence." Then the test begins. It is recorded how long it took the participant to complete the test.
Cognitive Dysfunction Evaluation - Serial Punctuation Test | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  SPT is a neurophysiological test that evaluates the neuromuscular system and motor control. It measures speed similarly to the LDT. The participant is given the page containing the SPT. "In this test, you are asked to put a dot in the middle of the round boxes. The point you need to pay attention to is not to skip the circles and when the line ends, continue from the left on the next line." It is recorded how many seconds the participant takes to complete the test.
Cognitive Dysfunction Evaluation - Line Drawing Test | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  LDT, like SPT, is a test that measures motor control and speed. The participant is given the page containing the LDT. "In this test, what is required of you is to draw a path with a pencil without extending between the two lines. The point you need to pay attention to is to continue throughout the entire page without raising your hand and when you make a mistake, do not go back and try to correct it." In this test, unlike the others, both how many seconds the participants took to complete the test and how many mistakes they made are recorded as two separate parameters.

SECONDARY OUTCOMES:
Muscle Strength | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  Participants' muscle strength will be evaluated by manual muscle test and hand grip strength test. Baseline® Hand Dynamometer (Fabrication Enterprises Inc., NY, USA), which is a valid and reliable dynamometer, will be used in manual muscle test. Baseline® Hydraulic Hand Dynamometer (Fabrication Enterprises Inc., NY, USA), which is also a valid and reliable dynamometer, will be used to evaluate hand grip strength test. In the manual muscle test, the Quadriceps muscle, one of the antigravity muscles, will be evaluated. Participants will be asked to maintain voluntary isometric contraction for 5 seconds and the value will be recorded in kilograms. Measurements will be repeated 3 times and a 1-minute rest period will be given between each measurement and the average of 3 measurements will be recorded. Hand grip strength measurement will be performed in the sitting position, which is the standard position recommended by the American Association of Hand Therapists, with the shoulder in addu
Muscle Mass | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  In the study published by Kara et al., it was reported that the cross-sectional area of the Quadriceps muscle was the average of the whole body. There is evidence that quadriceps muscle thickness is reduced in sarcopenic individuals. It has been emphasized that magnetic resonance imaging (MRI) and computed tomography (CT) imaging methods are superior to ultrasonography (US) imaging methods, but they have disadvantages in clinical use. US imaging method also has advantages. US imaging method is an easy, fast, safe, portable, valid (ICC: 0.92 - 0.99) and reliable (ICC: 0.88 - 0.97) alternative for measuring quadriceps muscle thickness. In our study, the muscle mass of the participants will be analyzed by evaluating the quadriceps muscle thickness with US imaging method.
Functionality - 6 Minute Walk Test | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  In the test, the maximum walking distance within 6 minutes is evaluated. During the test, the responses of systems such as the pulmonary and cardiovascular system, systemic circulation, peripheral circulation, neuromuscular structures and muscle metabolism are generally evaluated. Participants will be asked to walk as much distance as possible along a 30-meter corridor at their maximum speed, without running or jumping. All participants will be informed about the test, the application of the test and symptoms such as palpitations, shortness of breath and sweating that may occur during the test will be mentioned. The participants will be informed that they can leave the test at any time. A wheelchair will be available in the corridor. Participants will be allowed to rest on the chair at the starting line before starting the test. The time will start as soon participants start walking. Participants will not be allowed to talk off-topic during the test. Participants will be told to stop
Functionality - 5 Times Sit and Stand Test | Baseline, after 8th week, after 12th week, 6 months follow-up, 12 months follow-up
  The 5TSST was developed to measure functional lower extremity strength or to determine the movement strategies the participant uses to complete transfer skills. It is a test that measures how quickly one can move from sitting to standing 5 times in a row without using the upper extremities. In this test, participants will be seated in an armless chair, crossing their arms over their chest and without leaning their back on the backrest of the chair. The participant will be asked to sit down and stand up 5 times when "start" is said, and the stopwatch will be stopped when the participant sits on the chair for the fifth time. The test will be repeated twice, the first as practice, and the second measurement will be included in the statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, Study Director — Bahcesehir University, Department of Physiotherapy and Rehabilitation; Mustafa Oğuz Kethüdaoğlu, Principal Investigator — Sivas Cumhuriyet University,Department of Physiotherapy and Rehabilitation // Bahçeşehir University, Doctorate Program of Physiotherapy and Rehabilitation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal information will not be shared in accordance with the participant privacy and personal data protection law.